CLINICAL TRIAL: NCT02111031
Title: Registry to Demonstrate the Clinical Utility of CELLSEARCH® Circulating Tumor Cell (CTC) Test in Medicare-Eligible Metastatic Breast Cancer Patients
Brief Title: Clinical Utility of CTC Test in Medicare-Eligible Metastatic Breast Cancer Patients
Status: Withdrawn | Type: Observational
Why Stopped: The company decided not to start the study.
Sponsor: Janssen Diagnostics, LLC (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: JDX-2014-001
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Metastatic Breast Cancer; Breast Cancer
Keywords: CELLSEARCH; CTC; metastatic breast cancer; Registry; mBC
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Case: Patients with documented (histologically/pathologically confirmed) mBC diagnosis, at lease 65 years of age at documented mBC diagnosis, and actively treated by a physician at a participating cancer center who routinely (i.e., test at lease every quarter) use CTC testing (excluding patients who sought consults or second opinions).

SUMMARY:
The objective of the registry study is to demonstrate the clinical utility of the CELLSEARCH® CTC Test among the Medicare-Eligible metastatic Breast Cancer (mBC) patients in the United States. The objective of the present registry is to demonstrate the impact on patient management of the CELLSEARCH® CTC Test among the Medicare-eligible mBC patients. Hereto the hypothesis that the availability of CTC information provides clinicians important, timely information and impacts treatment decisions, will be tested.

This study is IDE-exempt since CELLSEARCH® CTC Test is a legally marketed device in the US, and is being used in accordance with its labeling.

ELIGIBILITY:
Inclusion Criteria:

Patient has documented (histologically/pathologically confirmed) mBC diagnosis

* Patient is at least 65 years of age at time of mBC diagnosis
* Patient is male or female
* Patient is being actively treated at the cancer center by a physician who uses or plans to use CTC testing on his mBC patients at lease every quarter.

Exclusion Criteria:

* Patients breast cancer is secondary not primary

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: "Cases" of CTC-tested mBC patients being cared for by physicians who routinely (i.e., test at least once every quarter) incorporate CTC testing in their management of mBC patients.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of treatment decisions that are indicated to be changed by the availability CTC results, stratified by relevant criteria (e.g. patient and tumor characteristics, concordance and discordance with other test results) | 15 months
  Percentage of treatment decisions that are indicated to be changed by the availability CTC results, stratified by relevant criteria (e.g. patient and tumor characteristics, concordance and discordance with other test results).
The percentage of treatment decisions for which CTC results are indicated to add value to treatment decision making, stratified by relevant criteria (e.g. patient and tumor characteristics, concordance and discordance with other test results) | 15 Months
  The percentage of treatment decisions for which CTC results are indicated to add value to treatment decision making, stratified by relevant criteria (e.g. patient and tumor characteristics, concordance and discordance with other test results)

SECONDARY OUTCOMES:
The relative value of CTC testing in treatment decisions as compared to other parameters, stratified by relevant criteria (e.g. patient and tumor characteristics, concordance and discordance with other test results) | 15 months
  The relative value of CTC testing in treatment decisions as compared to other parameters, stratified by relevant criteria (e.g. patient and tumor characteristics, concordance and discordance with other test results)
Overall survival, calculated as the median (+/- standard deviation [SD]) length of time from initial diagnosis to death. | 60 months
  Overall survival, calculated as the median (+/- standard deviation [SD]) length of time from initial diagnosis to death.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Montero, MD, Principal Investigator — Cleveland Clinic Main Campus
Locations (2):
- United States (2):
  - Abramson Cancer Center, University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania